CLINICAL TRIAL: NCT06119607
Title: A Prospective, Single-arm, Exploratory Clinical Investigation to Assess Preliminary Safety and Collect Performance and Effectiveness Data of the TRIFLO Heart Valve
Brief Title: PILot Aortic Triflo Valve Study
Acronym: PILATUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novostia SA (Industry)
Collaborators: Veranex (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100144; CIV-LT-23-08-043783 (Other: VASPVT)
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TRIFLO (Experimental)
  Interventions: Device: TRIFLO Heart Valve

INTERVENTIONS:
Device: TRIFLO Heart Valve — Surgical Aortic Valve Replacement - Mechanical Valve

SUMMARY:
A prospective, single arm, exploratory clinical investigation to assess preliminary safety and collect performance and effectiveness data of the TRIFLO Heart Valve.

DETAILED DESCRIPTION:
Up to 10 Subjects requiring aortic valve replacement of the native valve will be included in this First in Human clinical investigation on the TRIFLO Heart Valve device in Europe. The study is prospective, single-arm-open-label-non-randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 75 years old.
* Patient with symptomatic aortic valve disease (stenosis and/or regurgitation) where aortic valve replacement with a mechanical valve is recommended according to the decision of the site heart team and validated by the independent clinical review committee.
* Patient with a low surgical mortality risk with EuroSCORE II < 4%.
* Patient with echocardiographic Left Ventricular Ejection Fraction (LVEF) > 35% using Transthoracic Echocardiogram (TTE).
* Assessment using echocardiography imaging modality of annular suitable for a valve of 21 mm in size and acceptable for the Body Surface Area (BSA) of the patient to avoid any patient prosthesis mismatch.
* Participants are able to take low-dose aspirin at a dose of 75 -100 mg daily or have a documented contraindication to aspirin use.
* Patient is geographically stable and willing to return to implanting site for follow-up visits up to 5 years.
* Patient has been adequately informed of risks and requirements of the clinical investigation and is willing and able to provide informed consent for participation.
* In opinion of the Investigator, the patient has a life expectancy of at least 5 years.

Exclusion Criteria:

* Patient has a pre-existing prosthetic valve (including TAVI) or annuloplasty device or requires replacement or repair of the mitral, pulmonary or tricuspid valve.
* Patient is maintained on any permanent or long-term anticoagulant therapy (i.e. any A-fib, deep vein thrombosis, lung embolism, percutaneous coronary intervention (PCI), previous ST-elevation myocardial infarct (STEMI)).
* Patient has a history of vascular-related neurological events (TIA, stroke, intracranial bleeding) occurring within 6 months prior to enrollment.
* Patient has active endocarditis/myocarditis or other systemic infection within 3 months of the scheduled surgery.
* Patient has an additional cardiovascular pathology which would increase surgical risk of morbidity or mortality.
* Patient is planning another unrelated surgical procedure outside of the cardiac area within the next 12 months of study device implantation.
* Patient has renal insufficiency as determined by creatinine (S-Cr) level as ≥ 1.5 mg/dL or end stage renal disease requiring chronic dialysis at screening visit.
* Patient presents hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to planned valve surgery.
* Patient has active, clinically relevant bleeding disorder (documented leukopenia (WBC < 4.0 x 103/μL), acute anemia (Hgb < 10.0 g/dL or 6 mmol/L), thrombocytopenia (platelet count < 100 x 103/μL) or history of bleeding diathesis or coagulopathy).
* Patient has had prior organ transplant or is currently an organ transplant candidate.
* Patient is currently participating or participated in the last 30 days in another investigational device or drug trial.
* Patient who is pregnant, plan to become pregnant during the time of the clinical trial or is lactating or patient of childbearing age not taking any effective method of birth control.
* Patient is considered part of vulnerable population (i.e. prison inmates).
* Patient with documented history of substance (drug or alcohol) abuse within the last 5 years prior to implantation procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Safety - Mortality | At 12 and 18 months post procedure
  Rate of occurrence of all-cause mortality, cardiovascular, non-cardiovascular, and device-related mortality
Safety - Thrombotic events | Between 3 to 18 months post procedure
  Rate of valve related thrombotic events

SECONDARY OUTCOMES:
Safety - Major adverse cardiovascular events | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months
  Rate of occurrence of MACEs
Safety - Thromboembolism events | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months.
  Rate of occurrence of Transient Ischemic Attack (TIA), coronary and/or peripheral embolism
Safety - Thrombotic events | 24, 36, 48 and 60 months.
  Rate of valve-related thrombotic events
Safety - Atrial Fibrillation | 3, 9, 12, 15, 18, 24, 36, 48 and 60 months
  Rate of occurrence of New Onset Atrial Fibrillation
Safety - Endocarditis | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months.
  Rate of occurrence of Endocarditis
Safety - Hemolysis | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months.
  Rate of occurrence of Hemolysis followed by Plasma free hemoglobin
Safety - Reoperation | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months.
  Rate of occurrence of Reoperation
Safety - Structural & Non structural Valve Dysfunction | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months.
  Rate of occurrence of Structural & Non structural Valve Dysfunction
Safety - Bleeding | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months.
  Rate of occurrence of bleeding classified according to BARC
Safety - Pacemaker | 3 months
  Rate of occurrence New pacemaker implantation due to intervention
Safety - All-cause mortality | 1, 3, 9, 15, 24, 36, 48 and 60 months
  Rate of occurrence of All-cause mortality, cardiovascular, non-cardiovascular, and device related mortality
Safety - Procedural mortality | 1 month.
  Rate of occurrence of Procedural mortality
Performance - Procedure | Procedure
  Rate of initial success, correct positioning of a single TRIFLO Heart Valve into the proper anatomical location.
Performance - Hemodynamics | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months
  Change of hemodynamics compared to baseline followed by mean aortic valve pressure gradient
Performance - Regurgitation | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months
  Change of regurgitation class (As per VARC 3 Classification Guidelines) compared to baseline
Performance - EOA | 1, 3, 9, 12, 15, 18, 24, 36, 48 and 60 months
  Change of Effective Orifice Area (EOA) compared to baseline
Performance - Noise | 3, 9, 12, 15, 18, 24, 36, 48 and 60 months
  Assessment of noise perception - patient survey
Effectiveness - NYHA | 1, 3, 9, 12, 18, 24, 36, 48 and 60 months
  Change of NYHA Score compared to baseline
Effectiveness - QoL | 1, 3, 9, 12, 18, 24, 36, 48 and 60 months
  Change of Quality-of-life Score using KCCQ-12 questionnaires, compared to baseline
Effectiveness - 6MWT | 3, 9, 12, 18, 24, 36, 48 and 60 months
  Functional Assessment in 6-min walk test
Usability | Procedure
  Assessment of device handling ease by the physician - survey

CONTACTS AND LOCATIONS:
Overall Officials: Kęstutis Ručinskas, Prof., Principal Investigator — Vilnius University Hospital Santaros Clinics
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Vilnius County, Lithuania

IPD SHARING:
Plan to Share IPD: No